CLINICAL TRIAL: NCT01907633
Title: Post-Authorization Safety Study: Risk of Out-of-Hospital Sudden Cardiac Death in Users of Domperidone, Users of Proton Pump Inhibitors, and Users of Metoclopramide
Brief Title: An Observational Study to Assess the Risk of Out-of-Hospital Sudden Cardiac Death in Users of Domperidone, Users of Proton Pump Inhibitors, and Users of Metoclopramide
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR102051; RRA-7880 (Other: Janssen Research & Development, LLC); Epi 316 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Death, Sudden, Cardiac
Keywords: Death, Sudden, Cardiac; Risk of Sudden Cardiac Death; Domperidone; Proton Pump Inhibitors (PPI); Metoclopramide; Observational Study
MeSH Terms: conditions — Death, Sudden, Cardiac | interventions — Domperidone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Domperidone/ a proton pump inhibitor/metoclopramide users: Study patients had at least one prescription for domperidone, a proton pump inhibitor, or metoclopramide. Proton pump inhibitors observed in this study are: omeprazole, lansoprazole, esomeprazole, rabeprazole, and pantoprazole.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational and a retrospective study of existing data, so there will be no interventions. The exposure groups will be domperidone, proton pump inhibitors (omeprazole, lansoprazole, esomeprazole, rabeprazole, and pantoprazole), and metoclopramide.
  Other Names: Motilium

SUMMARY:
The purpose of this observational study is to assess the risk of out-of-hospital Sudden Cardiac (heart) Death (SCD) associated with current use of domperidone compared to current use of a Proton Pump Inhibitor (PPI), current use of metoclopramide, or non-use of any of these medications.

DETAILED DESCRIPTION:
This is a population-based, retrospective (a study in which the exposures and outcomes occurred before the study began), and nested case-control study (a study in which the patients with the study outcome [cases] and comparison patients without that outcome [controls] are observed to assess their exposure to the medication being studied [domperidone, PPI's and metoclopramide]). The data will come from the United Kingdom's Clinical Practice Research Datalink. The study will estimate the rate of SCD during periods of exposure to each of the study medications, and during periods of exposure to none of them; and the ratios of these rates. It will also use a "case-crossover" analysis (in which each case serves as his/her own control) to re-estimate these rate ratios in a manner that takes account of personal characteristics such as obesity or smoking that may affect the study findings and are incompletely recorded in the database.

ELIGIBILITY:
Inclusion criteria:

- Patients registered in English practices whose data are linkable to Hospital Episode Statistics (HES) and Office for National Statistics, UK (ONS). Patients are required to have at least 1 year in the Clinical Practice Research Datalink before they can enter the study

Exclusion criteria:

* Patients with a diagnosis of cancer other than non-melanoma skin cancer
* Patients from practices not linkable to HES and ONS data
* Patient time corresponding to the period between hospital admission date and 30 days after discharge date

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with exposure to domperidone, proton pump inhibitor, and metoclopramide
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of out-of-hospital sudden cardiac death (SCD) associated with the exposure to domperidone, proton pump inhibitor, metoclopramide, and none of these medications | 7 years
  This will be evaluated for the number of study participants (who had SCD) exposed to domperidone, proton pump inhibitor, metoclopramide, and none of these medications. SCD is defined as a natural death from an unexpected circulatory arrest, usually due to a cardiac arrhythmia (irregular heartbeat).
Number of out-of-hospital Sudden Cardiac Death (SCD) in relation to domperidone exposure period and domperidone non-exposure period | 7 years
  This will be evaluated for the number of study participants who had SCD in relation to domperidone exposure period and domperidone non-exposure period. SCD is defined as a natural death from an unexpected circulatory arrest, usually due to a cardiac arrhythmia (irregular heartbeat). This will be analyzed by case-crossover method (self-matching design) which will be adjusted for personal characteristics that vary little over time in each individual. eg, for obesity.
Number of out-of-hospital Sudden Cardiac Deaths (SCD) in relation to Proton Pump Inhibitor (PPI) exposure period and PPI non-exposure period | 7 years
  This will be evaluated for the number of study participants who had SCD in relation to PPI exposure period and PPI non-exposure period. SCD is defined as a natural death from an unexpected circulatory arrest, usually due to a cardiac arrhythmia (irregular heartbeat). This will be analyzed by case-crossover method (self-matching design) which will be adjusted for personal characteristics that vary little over time in each individual. eg, for obesity.
Number of out-of-hospital Sudden Cardiac Deaths (SCD) in relation to metoclopramide exposure period and metoclopramide non-exposure period | 7 years
  This will be evaluated for the number of study participants who had SCD in relation to metoclopramide exposure period and metoclopramide non-exposure period. SCD is defined as a natural death from an unexpected circulatory arrest, usually due to a cardiac arrhythmia (irregular heartbeat). This will be analyzed by case-crossover method (self-matching design) which will be adjusted for personal characteristics that vary little over time in each individual. eg, for obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC